CLINICAL TRIAL: NCT05985135
Title: Impact of Insulin Deprivation and Hyperglycemia on Plasma Protein Synthesis in People With Type 1 Diabetes Mellitus and Diabetes After Total Pancreatectomy
Brief Title: Impact of Insulin Deprivation and Hyperglycemia on Plasma Protein Synthesis in People With Type 1 Diabetes Mellitus
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, K. Sreekumaran Nair, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 21-000001
Record Dates: First submitted 2023-08-02; First posted 2023-08-14 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-01

CONDITIONS: Type 1 Diabetes
Keywords: Continuous subcutaneous insulin infusion; Multiple daily injections of insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Gels; Amino Acids; Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Type 1 Diabetes Mellitus (T1DM) Insulin Deprived (Experimental): Subjects will have their insulin infusions replaced with saline and have blood draws to monitor glucose levels along with a muscle biopsy following consumption of a Jell-O with Amino acids.
  Interventions: Procedure: Muscle Biopsy; Other: Jell-O with Amino acids
- Type 1 Diabetes Mellitus (T1DM) Insulin Treated (Experimental): Subjects will continue their baseline insulin infusion while maintaining a target blood glucose range. Blood draws will be obtained to monitor glucose levels along with a muscle biopsy following consumption of a Jell-O with Amino acids.
  Interventions: Procedure: Muscle Biopsy; Other: Jell-O with Amino acids
- Type 1 Diabetes Mellitus (T1DM) Insulin-Treated with Hyperglycemia (Experimental): Subjects will be continue their baseline insulin infusion for 2 hours and then receive an intravenous dextrose infusion to maintain elevated blood sugar levels. Blood draws will be obtained to monitor glucose levels along with a muscle biopsy following consumption of a Jell-O with Amino acids.
  Interventions: Procedure: Muscle Biopsy; Other: Jell-O with Amino acids; Dietary Supplement: Dextrose
- Non-Diabetic Controls (Other): Subjects will have blood draws to monitor glucose levels along with a muscle biopsy following consumption of a Jell-O with Amino acids.
  Interventions: Procedure: Muscle Biopsy; Other: Jell-O with Amino acids
- Diabetes after Total Pancreatectomized (DATP) Insulin Treated (Experimental): Subjects will continue their baseline insulin infusion while maintaining a target blood glucose range. Blood draws will be obtained to monitor glucose levels along with a muscle biopsy following consumption of a Jell-O with Amino acids.
  Interventions: Procedure: Muscle Biopsy; Other: Jell-O with Amino acids
- Diabetes after Total Pancreatectomized (DATP) Insulin Deprived (Experimental): Subjects will have their insulin infusions replaced with saline and have blood draws to monitor glucose levels along with a muscle biopsy following consumption of a Jell-O with Amino acids.
  Interventions: Procedure: Muscle Biopsy; Other: Jell-O with Amino acids

INTERVENTIONS:
Procedure: Muscle Biopsy — Needle muscle biopsy of the outer thigh muscle
Other: Jell-O with Amino acids — An amino acid mixture containing 13C6 Lysine isotope label
Dietary Supplement: Dextrose — Intravenous form of sugar
  Arms: Type 1 Diabetes Mellitus (T1DM) Insulin-Treated with Hyperglycemia

SUMMARY:
This research is being done to better understand how insulin effects muscle, blood, and the body in people with Type 1 Diabetes.

DETAILED DESCRIPTION:
Insulin's contribution in controlling glucose homeostasis has been well appreciated but, its role in maintaining proteome homeostasis is less understood. Some animal and human studies have demonstrated that insulin signaling regulates protein synthesis and degradation as well as posttranslational modifications at the tissue level. Insulin's effect on the muscle's mitochondrial proteo-stasis has also been elucidated. Insulin deprivation increases global synthesis of splanchnic proteins based on isotope dilution studies across splanchnic bed. Most plasma proteins are derived from liver and preliminary studies suggest that synthesis rates of some plasma proteins increase while others decrease. Fractional rates of synthesis of various plasma proteins from the liver have been demonstrated in insulin deprivation state. These proteins might be implicated in the development of some of the complications from diabetes mellitus type 1. (T1DM) especially of macrovascular. Researchers have recently developed an isotope-based methodology to simultaneously measure in vivo synthesis rates of multiple plasma proteins in human.

In order to further investigate the effects of insulin deprivation researchers will apply the novel non-radioactive stable isotope-based approach on the rate of different plasma protein synthesis in T1DM and Diabetes after total pancreatectomy (DATP) in comparison with non-diabetic controls. Researchers will study pancreatectomized people because like T1DM they also are insulin deficient but unlike pancreatectomized people also are deficient in glucagon. Some tantalizing data from many studies indicate that glucagon also have catabolic effect not only on liver derived proteins but also on skeletal muscle-based proteins. Since skeletal muscle has no glucagon receptors, researchers hypothesize that unknown factors are released to the circulation that act on skeletal muscle to release amino acids for consumption in liver. Researchers will measure amino metabolites, acyl carnitines, organic acids, and ceramides in plasma and determine the blood exosome cargo by mass spectrometry-proteins and lipids and miRNA by PCR.

Researchers have previously shown reduced muscle mitochondrial ATP production during insulin deprivation in both T1D humans and diabetic mice and here researchers will measure mitochondrial energy dynamics in all study participants by the established techniques available in our lab.

ELIGIBILITY:
Inclusion Criteria - Type 1 Diabetes Group:

- Able to provide written consent.

Exclusion Criteria - Type 1 Diabetes Group::

* BMI < 20 or > 32 kg/m^2.
* Celiac disease.
* Pregnancy.
* Smoking.
* Reported history of illicit substance use.
* History of active cardiovascular, cerebrovascular, or peripheral vascular disease.
* Active renal disease evidenced by estimated glomerular filtration rate (GFR) < 50 mL/min/1.73 m^2.
* Severe peripheral or autonomic neuropathy.
* Dementia or any other neurologic disease.
* Uncontrolled psychiatric disease.
* Any learning disability.
* Anemia.
* Thyroid-stimulating hormone (TSH) ≥ 7 or TSH ≤ 7 and free T4 ≤ 0.9.
* Hemoglobin A1c > 9.0%.
* Type 2 Diabetes Mellitus (T2DM), or impaired fasting glucose.
* Detectable C peptide.

Inclusion Criteria - Control Group:

* Able to provide written consent.
* T1DM treated with continuous subcutaneous insulin infusion (CSII) or multiple daily injections (MDI) (not Degludec).

Exclusion Criteria - Control Group:

* BMI < 20 or > 32 kg/m^2.
* Celiac disease.
* Pregnancy.
* Smoking.
* Reported history of illicit substance use.
* History of active cardiovascular, cerebrovascular, or peripheral vascular disease.
* Active renal disease evidenced by estimated GFR < 50 mL/min/1.73 m^2.
* Severe peripheral or autonomic neuropathy.
* Dementia or any other neurologic disease.
* Uncontrolled psychiatric disease.
* Any learning disability.
* Anemia.
* TSH ≥ 7 or TSH ≤ 7 and free T4 ≤ 0.9.
* T2DM, or impaired fasting glucose.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Protein synthesis | Approximately 7 hours
  Measurement of isotope abundance in peptides derived from the digested proteins

CONTACTS AND LOCATIONS:
Overall Officials: K. Sreekumaran Nair, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials